CLINICAL TRIAL: NCT04763655
Title: Neural Biomarkers of Electroconvulsive Therapy Response in Schizophrenia
Brief Title: Neural Biomarkers of Electroconvulsive Therapy Response
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0100; K23MH120504 (NIH)
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Electroconvulsive Therapy Treated Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment as usual (Other)
  Interventions: Diagnostic Test: clinical and neuropsychological testing

INTERVENTIONS:
Diagnostic Test: clinical and neuropsychological testing — Patients are monitored with Brief Psychiatric Rating Scale (BPRS) weekly and structural and functional MRI and MATRICS battery before and at the end of the course of the study
  Other Names: MRI of the brain

SUMMARY:
In the proposed study, the investigators will utilize resting-state functional MRI (fMRI) and structural MRI-based electrical field modeling to study the effect of electroconvulsive therapy on human neural circuitry. Our study will recruit patients who are beginning treatment with bilateral electroconvulsive therapy (N=75). Our design will be longitudinal where patients will be followed up until their 8th week electroconvulsive therapy clinically. The primary measure of interest will be the slope of clinical change estimated with mixed effect modeling (see Approach). Secondary measures will be the cognitive performance change between baseline and the 8th week electroconvulsive therapy time point.

ELIGIBILITY:
Inclusion Criteria:

1. current positive symptoms rated ≥4 (moderate) on one or more of these BPRS 53 items: hallucinatory behavior, unusual thought content, suspiciousness, conceptual disorganization;
2. has failed at least one trial of treatment with antipsychotic drug, lasting 6 weeks in duration,
3. competent and willing to sign informed consent;
4. for women, negative pregnancy test and agreement to use a medically accepted birth control method; and
5. Diagnostic and Statistical Manual (DSM)-IV diagnosis of schizophrenia, schizoaffective or schizophreniform disorder.

Exclusion Criteria:

1. serious neurological or endocrine disorder;
2. any medical condition which requires treatment with a medication with psychotropic effects;
3. significant risk of suicidal or homicidal behavior;
4. cognitive (MMSE ≤ 23) or language limitations that would preclude subjects providing informed consent;
5. contraindications to treatment with electroconvulsive therapy;
6. contraindications to magnetic resonance imaging (e.g. pacemaker)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Response to Brief Psychiatry Rating Scale (BPRS) | Baseline and 8 weeks.
  The change of total BPRS score between Week 8 and Baseline divided by baseline (percentage change). The change in the total score which can be between 18-126 (in extreme cases) will be reported.

SECONDARY OUTCOMES:
The change of the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) | Baseline and 8 weeks.
  Using the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) neuropsychology battery, the age corrected standardized total T-scores change will be reported.
Volume change of the hippocampus bilaterally based on MRI based volumetry | Baseline and 8 weeks.
  Volume change in the hippocampus measured by subtracting the volume of the bilateral hippocampus at 8th week from baseline divided by baseline (percentage). A longitudinal FreeSurfer (MGH) will be used to measure the volumes of the hippocampus in cubic centimeters and the change will be reported.
Magnitude of the electric field in the hippocampus bilaterally | At baseline.
  The electrical field will be estimated with finite element modeling from the structural scans in the hippocampus (Volt per meter). A Matlab based program called ROAST (developed at CUNY) to estimate the electric field in the hippocampus and the average electric field magnitude across the hippocampus will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Argyelan, MD, Principal Investigator — The Zucker Hillside Hospital
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is shared via the National Institute of Mental Health Data Archive mechanisms.